CLINICAL TRIAL: NCT02068976
Title: Observational Epidemiologic Study in Women With Premature Ovarian Failure (POF)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-IOP-2012-109
Record Dates: First submitted 2014-02-17; First posted 2014-02-21 (Estimated); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Primary Ovarian Insufficiency
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women with Primary Ovarian Insufficiency

SUMMARY:
This is an observational epidemiologic multicentric study of follow-up a cohort for described the situation of patients with primary ovarian insufficiency in public population with respect to the age of apparition the primary ovarian insufficiency .

iPOI (Investigators in premature ovarian insufficiency): M. Guinot, B. Roca, J. Tomás, P. Escamilla, J. Hernández, P. Llaneza, N. Mendoza Ladrón de Guevara, B. Otero García, I. Ñiguez, A. Castro, L. Baquedano, P. Romero, S. Sánchez.

ELIGIBILITY:
Inclusion criteria:

* Women between 18 years and 39 years.
* Primary ovarian insufficiency demonstrated with amenorrhea and levels of follicle stimulating hormone (FSH) over to 40 IU in two determinations measured with a difference of one moth.
* Not present linguistic barriers ,shaw attitude towards collaboration ,be able to attend the study center for all follow-up visits.
* Signed informed consent before inclusion in the study and after having been informed of the procedures performed in this study.

Exclusion criteria :

* Women with secondary hormonal alteration that do no meet the diagnostic criteria of the disease.
* Refusal to participate.
* Withdrawal of informed consent.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients procedints of gynecology deparment of the centers participants
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-11-28 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Age | Day 0
  Age when diagnosed primary ovarian insufficiency

CONTACTS AND LOCATIONS:
Overall Officials: Misericordia Guinot, MD PhD, Study Chair — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (15):
- Spain (15):
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Hospital Universitario Materno Infantil de Canarias, Las Palmas de Gran Canaria, Las Palmas
  - Hospital de Manacor, Manacor, Palma de Mallorca
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital de Poniente de El Egido, Almería
  - Complejo Asistencial de Avila, Ávila
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Terrasa, Barcelona
  - Hospital Universitari Mutua de Terrasa, Barcelona
  - Hospital Universitario de Cruces, Bilbao
  - Hospital Universitario Virgen de las Nieves, Granada
  - Universidad de Granada, Granada
  - Grupo Hospitalario Perpetuo Socorro, Lleida
  - HCU Virgen de la Arrixaca, Murcia
  - Hospital Universitario Miguel Servet, Zaragoza